CLINICAL TRIAL: NCT00203788
Title: Developmental Processes in Schizophrenic Disorders: Improving and Predicting Work Outcome in Recent-Onset Schizophrenia
Brief Title: Improving Work Outcome in People With Recent-onset Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Keith Nuechterlein, Ph.D., Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH037705 (NIH); R01MH037705 (NIH); Janssen RIS-USA-67; DAHBR AD-P
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2008-05

CONDITIONS: Schizophrenia
Keywords: work outcome; supported employment; social skills training; risperidone; cognition; first-episode schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Palliative Care; Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Individual Placement and Support Plus Workplace Fundamentals Module
  Interventions: Behavioral: Individual Placement and Support; Behavioral: Workplace Fundamentals Module; Drug: Oral risperidone
- 2 (Active Comparator): Brokered Vocational Rehabilitation
  Interventions: Behavioral: Brokered Vocational Rehabilitation; Drug: Oral risperidone; Behavioral: Skills training group

INTERVENTIONS:
Behavioral: Individual Placement and Support — Supported education/employment
  Arms: 1
Behavioral: Workplace Fundamentals Module — Group skills training on job/school topics
  Arms: 1
Behavioral: Brokered Vocational Rehabilitation — Vocational rehabilitation through traditional separate state-funded agency
  Arms: 2
Drug: Oral risperidone — Risperidone, starting target dosage was 6 mg, adjusted to level judged optimal by treating psychiatrist
  Other Names: Risperdal
Behavioral: Skills training group — Group social skills training that did not focus primarily on work situations
  Arms: 2

SUMMARY:
This study will determine the effectiveness of combining antipsychotic medication with Individual Placement and Support (IPS) and group training with the Workplace Fundamentals Module or Brokered Vocational Rehabilitation in facilitating the search for appropriate work or schooling and maintaining work or school activities in people with recent-onset schizophrenia.

DETAILED DESCRIPTION:
The purpose of this protocol is to test, in recent-onset schizophrenia, the efficacy of a rehabilitative intervention that is designed to enhance the search for appropriate work or schooling and to increase ability to maintain work or school activities more successfully. Predictors of work outcome are being assessed in the context of this work rehabilitation and treatment with the second-generation antipsychotic medication, risperidone.

The Developmental Processes in Schizophrenic Disorders project involves an ongoing series of longitudinal follow-through studies of individuals with a recent onset of schizophrenia. The current protocol focuses particularly on processes affecting work outcome in this initial period after onset of schizophrenia, drawing on findings that link cognitive deficits in schizophrenia to functional outcome. The protocol is determining the effects on work outcome of a rehabilitative intervention designed to enhance search for appropriate work or schooling and to increase ability to maintain work or school activities more successfully. All entering patients are placed on a common antipsychotic medication, oral risperidone, and are provided clinical treatment by a psychiatrist and a case manager. Participating patients are randomly assigned to a combination of Individual Placement and Support (IPS) and group training with the Workplace Fundamentals Module or to a Brokered Vocational Rehabilitation Model.

The protocol is examining the predictors of level of work functioning attained in the context of the work-focused intervention and maintenance on risperidone. Potential neurocognitive and environmental predictors of work and social functioning and clinical course are being examined. Aspects of early perceptual processing, allocation of attention, working memory, secondary verbal memory, and conceptual flexibility that are implicated as influences on functional outcome are assessed, as are potential stresses and supportive influences in the environment.

ELIGIBILITY:
Inclusion Criteria:

* First major psychotic episode within 2 years of study entry
* RDC schizophrenia or schizoaffective disorder, mainly schizophrenic subtype
* Residence within commuting distance of UCLA
* Interest in trying to resume work or school
* Speaks English

Exclusion Criteria:

* Known neurological disorder
* Significant and habitual drug abuse or alcoholism within 6 months of psychotic episode or evidence that substance abuse will be a prominent factor in course of illness
* Mental retardation
* Treatment with risperidone is contraindicated

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 1999-05; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Return to regular work or school during 18 month trial (SAS Work Section) | Every 3 months
Maintenance of work/school attendance over 18 months (SAS) | Every 3 months
Quality of work functioning on Work Behavior Inventory | Baseline, 6 months, 18 months

SECONDARY OUTCOMES:
Cognitive performance on test battery | Baseline, 6 months, 18 months
Exacerbation or relapse of psychotic symptoms (BPRS) | Every 2 weeks
Retention in treatment | Every 3 months
Awareness of illness (SUMD-R) | Entry, 6 months, 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Keith H Nuechterlein, PhD, Principal Investigator — University of California, Los Angeles, Department of Psychiatry and Biobehavioral Sciences
Locations (1):
- UCLA Neuropsychiatric Institute, Los Angeles, California, United States

REFERENCES:
- [Background] Nuechterlein KH, Subotnik KL, Ventura J, Gitlin MF, Green MF, Wallace CJ, Becker DR, Liberman RP, Drake RE, Mintz J. Advances in improving and predicting work outcome in recent-onset schizophrenia. Schizophrenia Bulletin 31(2): 530, 2005.